CLINICAL TRIAL: NCT07393997
Title: Clinical Evaluation of Autogenous Tooth Transplantation With Instrumentally Simulated Open Apex and Autologous Platelet-Rich Fibrin (PRF) Support in Teeth With Complete Root Formation
Brief Title: Autogenous Tooth Transplantation With Instrumentally Simulated Open Apex and Platelet-Rich Fibrin
Acronym: OpenApexT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bari Aldo Moro (Other)
Responsible Party: Principal Investigator, Giuseppe D'Albis, Principal Investigator, University of Bari Aldo Moro
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OpenApexTechnique
Record Dates: First submitted 2026-01-23; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Tooth Loss; Tooth Diseases; Reimplant; Complications
MeSH Terms: conditions — Tooth Loss; Tooth Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tooth loss (Experimental): Patients presenting with hopeless teeth
  Interventions: Procedure: Autogenous Tooth Transplantation; Procedure: Alveolar Prf graft

INTERVENTIONS:
Procedure: Autogenous Tooth Transplantation — After atraumatic extraction of the donor tooth, a simulated apical opening will be created using rotary instruments to induce apical patency and replicate the biological conditions of an open apex, potentially favoring pulpal revascularization.
Procedure: Alveolar Prf graft — To enhance clot formation and promote angiogenesis and tissue regeneration, autologous platelet-rich fibrin (PRF) will be used in the recipient site.
  PRF Collection and Preparation
  * Prior to surgery, peripheral venous blood will be collected from the patient using sterile tubes without anticoagulants.
  * The blood samples will be immediately processed using a standardized centrifugation protocol, allowing the separation of a fibrin matrix enriched with platelets and leukocytes.
  * After centrifugation, the PRF clot will be gently removed and prepared under sterile conditions for clinical use.
  PRF Placement
  * The autologous PRF will be placed directly into the recipient alveolus before positioning the donor tooth.
  * The PRF matrix will act as a biological scaffold, promoting clot stabilization, neovascularization, and early healing of the periodontal and pulpal tissues.

SUMMARY:
Autogenous tooth transplantation (autotransplantation) represents a biologically valid alternative to implant therapy, particularly in young patients where implant placement is contraindicated due to ongoing skeletal growth. This approach preserves alveolar bone volume, maintains periodontal proprioception, and allows physiological adaptation over time.

DETAILED DESCRIPTION:
One of the main limitations of autotransplantation in teeth with complete root formation is the absence of pulpal revascularization following apical closure, which frequently leads to pulp necrosis and the subsequent need for endodontic treatment. Root canal therapy may compromise the structural integrity of the tooth and negatively affect long-term outcomes.

The combined use of simulated apical patency and autologous PRF is expected to enhance pulpal revascularization, reduce the incidence of pulp necrosis, and improve the biological and clinical outcomes of autogenous tooth transplantation in teeth with complete root formation.

This protocol aims to expand the indications for autogenous tooth transplantation by introducing a biologically driven approach that combines surgical and regenerative techniques. The use of autologous PRF may represent a valuable adjunct in improving healing and long-term success in challenging clinical scenarios.

ELIGIBILITY:
Inclusion Criteria:

Autotransplantation will be performed in selected cases with favorable biological and functional prognosis, including:

* Early loss of permanent teeth due to trauma, extensive caries, or agenesis.
* Dental agenesis, particularly involving premolars or incisors, when a suitable donor tooth is available.
* Replacement of non-restorable teeth (fractures or destructive caries).
* Preservation of alveolar bone in growing patients where implant therapy is contraindicated.
* Functional and aesthetic rehabilitation of anterior teeth in pediatric and adolescent patients.
* Post-traumatic oral rehabilitation in young patients.
* Good general and oral health.
* Presence of a vital and intact periodontal ligament on the donor tooth.
* Adequate recipient site dimensions and morphology, or surgically adaptable.
* Absence of active infection at the recipient site. Donor Tooth Selection Criteria
* Tooth extracted for orthodontic purposes.
* Impacted or erupting third molars with compatible morphology.
* Suitable supernumerary teeth.

Exclusion Criteria:

* Poor patient compliance.
* Active infection at the recipient site.
* Smoking of more than 15 cigarettes a day

  •. Untreated periodontal disease
* Pregnancy or breastfeeding at date of inclusion
* Acute infections

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Resporption | 1 month, 3 months, 6 months, 1 year, 2 years
  Rx to evalue internal or external root resorption. Present or Not.
Vitality | 1 month, 3 months, 6 months, 1 year, 2 years
  Pulp vitality will be assessed during follow-up using standardized sensibility tests. ( electric test). Vitality : Yes or None
Mobility | 1 month, 3 months, 6 months, 1 year, 2 years
  Mobility Test. Grade I, Grade II or Grade III
Inflammation | 1 month, 3 months, 6 months, 1 year, 2 years
  signs of inflammation will be monitored. Blood on Probing: Yes or None
periodontal health | 1 month, 3 months, 6 months, 1 year, 2 years
  Periodontal Chart (mm). 6 point for each tooth.
bone remodeling | 1 month, 1 year, 2 years
  Assess periodontal integration and bone remodeling by Rx. Comparing Rx.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe D'Albis, Dr., Principal Investigator — University of Bari Aldo Moro; Nicola De Giglio, Dr., Principal Investigator — University of Bari Aldo Moro; Saverio Capodiferro, Prof. Dr., Study Director — University of Bari Aldo Moro
Locations (1):
- University of Bari Aldo Moro, Hospital, Bari, Italy